CLINICAL TRIAL: NCT06238336
Title: Clinical Study of CAR-T Technology for the Treatment of Relapsed Refractory Malignant Haematological Tumours
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-2019-114
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy (Experimental): Dose climbing started with 1.0*10^6/kg back infusion, 3 patients per dose group, if there is no adverse reaction the dose can be increased to 2.0*10^6/kg, 4.0*10^6/kg, the maximum dose can be extended the study.
  Interventions: Drug: CAR-T cell therapy

INTERVENTIONS:
Drug: CAR-T cell therapy — The application of CAR-T therapy in the clinic generally involves the in vitro preparation and in vivo infusion of CAR-T, and the specific experimental process is divided into five steps: (1) isolation of T cells from the peripheral blood of the cancer subjects or single harvested single nucleated cells; (2) use of genetic engineering to transfer CAR structural genes that can specifically recognise the tumour cells into the T cells; (3) in vitro cultivation and expansion of CAR-T cells to the desired infusion dose (4) Non-myeloablative chemotherapy is administered prior to the infusion of CAR-T cells, which is used to remove immunosuppressive cells and reduce the tumour load so as to enhance the efficacy of the treatment; (5) CAR-T cells are infused according to the expected dosage, and the efficacy of the treatment is observed and the adverse reactions are closely monitored.

SUMMARY:
The trial is designed as an early exploratory single-centre, open, single-arm clinical trial. The trial is planned to evaluate the safety and efficacy of CAR-T for the treatment of relapsed refractory malignant haematological tumours. The trial is divided into five visit periods as follows: screening period, non-myeloablative pretreatment, short-term follow-up period, mid-term follow-up period and exit visit.

DETAILED DESCRIPTION:
1) Screening period (-21 to -7 days, 2 weeks): subjects signed the informed consent form and completed a series of examinations, and it was judged by the investigator whether subjects met the inclusion criteria and did not meet the exclusion criteria based on the results of the examinations and the inclusion/exclusion criteria. And the investigator will judge whether some of the examination results within one month before the date of informed consent are acceptable according to the patient's condition.

2) Non-myeloablative preconditioning (-4 to -1 days for 4 days): the need for preconditioning and the preconditioning regimen were decided based on the subject's condition, and the most commonly used regimen was the FC regimen. After returning to the study centre for admission at the time notified by the investigator, subjects received fludarabine and cyclophosphamide on days -4 to -2 of the trial; the drugs were discontinued for 1 day on day -1 and a series of tests were completed as baseline information for subjects after non-clear myeloid preconditioning;

3) Short-term follow-up period (visits 4 to 10: 0 to 180 days over a period of 6 months): subjects return to the study centre for a series of examinations every month for 6 months following the start of infusing back the expected dose of CAR-T cells on Day 0 of the trial. The investigator evaluates the short-term safety and efficacy of CAR-T therapy based on the subjects' examination results;

4) Medium- to long-term follow-up period (180 to 360 days over a period of 6 months): subjects will return to the research centre every 2 months for a series of examinations within 6 months after completion of the short-term follow-up. The investigators will evaluate the mid- and long-term safety and efficacy of CAR-T therapy based on the subjects' examination results;

5) Withdrawal Visit (at any time): all subjects may withdraw from this study at any stage of the trial, with or without providing a reason. If the subject withdraws from the study after the return of the CAR-T cells, he/she will be required to complete the examination items required for the withdrawal visit in the visit flowchart; if the subject withdraws from the visit prior to the return of the CAR-T cells, he/she will be required to complete the safety examination items only, and the reason for the subject's withdrawal will be recorded in detail by the investigator. If the subject stops treatment due to AE, the investigator will follow the subject for necessary safety visits until the subject's AE returns to baseline levels or reaches steady state.

ELIGIBILITY:
Inclusion Criteria:

1. patients or their legal guardians voluntarily participate and sign an informed consent form;
2. male or female patients aged 14 to 70 years (inclusive);
3. be diagnosed as malignant haematological tumour by pathological and histological examination;
4. have a measurable or evaluable lesion;
5. the patient has good function of major tissues and organs:

(1) Liver function: ALT/AST <3 times upper limit of normal (ULN) and total bilirubin ≤34.2 μmol/L; (2) Renal function: creatinine <220 μmol/L; (3) Lung function: room oxygen saturation ≥95%; (4) Cardiac function: left ventricular ejection fraction (LVEF) ≥40%. (6) Patient's peripheral superficial venous blood flow is smooth and can meet the demand of intravenous drip; 7. patients with ECOG score ≤2 and expected survival time ≥3 months.

Exclusion Criteria:

1. Women who are pregnant (positive urine/blood pregnancy test) or breastfeeding;
2. men or women who are planning to conceive within the last 1 year;
3. patients who cannot guarantee effective contraception (condoms or birth control pills, etc.) within 1 year of enrolment;
4. patients with uncontrolled infections within 4 weeks prior to enrolment;
5. active viral hepatitis B/C;
6. patients with HIV infection;
7. patients with severe autoimmune diseases or immunodeficiency diseases;
8. patients who are allergic to large molecule biopharmaceuticals such as antibodies or cytokines;
9. patients who have participated in other clinical trials within 6 weeks prior to enrolment;
10. the patient has used hormones systematically within 4 weeks prior to enrolment (except for patients using inhaled hormones);
11. the patient has a psychiatric disorder
12. the patient has substance abuse/addiction;
13. other conditions that, in the judgement of the investigator, make the patient unsuitable for enrolment.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 36 months
  Adverse events associated with CAR-T therapy, serious adverse events and clinically significant laboratory test abnormalities.

SECONDARY OUTCOMES:
CAR-T amplification levels | Up to 36 months
  Characterisation of CAR-T cell expansion levels in subjects (peripheral blood, bone marrow, cerebrospinal fluid and lymph nodes, etc.) over time.
Duration of the CAR-T | Up to 36 months
  Duration of CAR-T cell persistence in subjects (peripheral blood, bone marrow, cerebrospinal fluid and lymph nodes, etc.
Lymphocyte abatement | Up to 36 months
  The characteristics of lymphocyte ablation in the subject.
Objective Response Rate (ORR) | Up to 6 months
  Proportion of patients whose tumour volume shrinks to a pre-specified value and who are able to maintain the minimum timeframe required, as the sum of the proportions in complete and partial remission. Objective tumour remission rates at 3 months, 6 months and 1 year follow-up after treatment.It is the sum of the proportions of complete remission (CR) and partial remission (PR).
Progression-free survival(PFS) | Up to 36 months
  Time from start of patient's treatment to disease progression or death from any cause
Event free survival (EFS) | Up to 36 months
  Time from the start of enrolment to the occurrence of any event.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomin Zhang, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- ShanxiBethuneH, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No